CLINICAL TRIAL: NCT01273701
Title: Combination of Psychosocial Intervention and Slow Prosecutions for the Treatment of Methamphetamine Abuse/Dependence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Yi-Ting, Lin/M.D., Department of Psychiatry, National Taiwan University Hospital Yunlin Branch
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201011014RB
Record Dates: First submitted 2011-01-06; First posted 2011-01-10 (Estimated); Last update posted 2011-01-10 (Estimated); Status verified 2010-12

CONDITIONS: Amphetamine Abuse; Amphetamine Dependence; Methamphetamine Abuse; Methamphetamine Dependence
Keywords: amphetamine; methamphetamine; psychosocial intervention; contingency management; slow prosecution; substance use disorder
MeSH Terms: conditions — Amphetamine-Related Disorders; Substance-Related Disorders | interventions — Psychosocial Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- TSTSU-N (Experimental): TSTSU-N stands for Treatment for Schedule Two Substance Use, No Telephone Reminding. Subjects will be referred by the Yunlin District Prosecutors Office for one-year psychosocial interventions to get slow prosecutions. After the referral, they will be randomized in a 1:1 ratio to either TSTSU-N group or TSTSU-T group. During the intervention, subjects of TSTSU-N will not receive telephone reminding before each visit.
  Interventions: Behavioral: Psychosocial intervention
- TSTSU-T (Experimental): TSTSU-T stands for Treatment for Schedule Two Substance Use, Telephone Reminding. Subjects will be referred by the Yunlin District Prosecutors Office for one-year psychosocial interventions to get slow prosecutions. After the referral, they will be randomized in a 1:1 ratio to either TSTSU-N group or TSTSU-T group. During the intervention, subjects of TSTSU-T will receive telephone reminding before each visit.
  Interventions: Behavioral: Psychosocial intervention; Behavioral: Telephone reminding
- OPD (Active Comparator): OPD stands for Outpatient Department. Subjects in this arm will be methamphetamine users who voluntarily visit psychiatric clinics for treatment of mental disorders in National Taiwan University Hospital, Yunlin Branch. They will be referred to this study by their treating psychiatrists.
  Interventions: Behavioral: Psychosocial intervention

INTERVENTIONS:
Behavioral: Psychosocial intervention — The treatment is one-year long and composed of 3 stages of psychosocial intervention. Subjects of TSTSU arms receive urine methamphetamine examinations at each visit, while subjects in OPD arm being tested at first/last visits and during stage changes.
  -Stage 1, early intensive monitoring stage: The visit interval is 1 week. If the urine tests and self-report on methamphetamine use are negative for consecutive 4 visits, subjects can proceed to stage 2. (In OPD arm, the visit interval can be 2 weeks according to subjects' requirements.)
  -Sage 2, late intensive monitoring stage: The visit interval is 2 week. If the urine tests and self-reports are straightly negative for 4 visits, subjects can proceed to stage 3. Whenever recent methamphetamine is detected, subjects should move back to stage 1.
  -Stage 3, usual monitoring stage: The visit interval is 1 month until the end of treatment. Whenever recent methamphetamine is detected, subjects should move back to stage 1.
  Other Names: Contingency management
Behavioral: Telephone reminding — Subjects in TSTSU-T group will receive addition telephone reminding one day before each visit. Each call will be no longer than five minutes. On the telephone, brief motivation enhancement may be conducted.
  Arms: TSTSU-T

SUMMARY:
The hospital where this study will be conducted is responsible for the one-year contingency management treatment for methamphetamine drug offenders referred from the Yunlin District Prosecutors Office. Completing the one-year treatment is prerequisite for offenders to get slow prosecutions.

It is an open-label, parallel-group trial comparing the combination of psychosocial intervention and slow prosecutions with psychosocial intervention alone in treating subjects with methamphetamine dependence

Study Hypothesis

1. Psychosocial interventions in combination with slow prosecutions is more effective than psychosocial interventions alone to achieve abstinence for subjects with methamphetamine abuse/dependance.
2. Inclusion of telephone reminding before each visit will enhance the retention rate and abstinence rate.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV-TR criteria for amphetamine/methamphetamine abuse or dependence
* 18 - 65 years old
* For TSTSU-N and TSTSU-T arms: methamphetamine offenders referred by the Yunlin District Prosecutors Office
* For OPD arm: psychiatric outpatients referred from the psychiatry clinics in National Taiwan University Hospital, Yunlin Branch

Exclusion Criteria:

* Concurrent use of other illicit substances
* Co-morbidity with major psychotic disorders (schizophrenia, schizoaffective disorder, other psychotic disorder), mental retardation, acute episodes of major depressive disorder or bipolar affective disorder) or serious personality disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Endpoint abstinence rate | At the end of one-year treatment
  According to the urine amphetamine/methamphetamine screen after the one-year treatment, negative result suggests successful abstinence.

SECONDARY OUTCOMES:
Retention rate | during the whole one-year treatment
  proportion of subjects who can complete the course of one-year treatment
Length of retention | during the whole one-year treatment
  the averaged duration of attending treatment
The longest period of abstinence | during the whole one-year treatment
  the longest period of time with successive negative results of urine amphetamine/methamphetamine tests or negative reports of recent methamphetamine use

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Ting Lin, M.D., Principal Investigator — Department of Psychiatry, National Taiwan University Hospital Yunlin Branch
Locations (1):
- National Taiwan University Hospital Yunlin Branch, Yunlin, Taiwan, Taiwan